CLINICAL TRIAL: NCT01932489
Title: THE JULES BORDET INSTITUTE PROGRAM FOR MOLECULAR PROFILING OF METASTATIC LESIONS: FEASIBILITY. PRECISION - Feasibility.
Brief Title: The Jules Bordet Institute Molecular Profiling Program Feasibility Trial
Acronym: PRECISION-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IJBCE2139
Record Dates: First submitted 2013-08-23; First posted 2013-08-30 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2014-10

CONDITIONS: Colorectal Cancer Metastatic; Metastatic Melanoma; Metastatic Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequencing of a metastatic lesion. (Other): Biopsy of a metastatic lesion followed by a targeted cancer gene screen.
  Interventions: Procedure: Biopsy of a metastatic lesion.

INTERVENTIONS:
Procedure: Biopsy of a metastatic lesion.

SUMMARY:
Prior to the use of genomic tests for patient inclusion in clinical trials, it is essential for the Jules Bordet Institute (JBI) to pilot the logistical and technical aspects by examining the feasibility and turnaround time of performing and obtaining data from a few key molecular assays.

Patients with metastatic colorectal cancer, non-small cell lung cancer or melanoma will be enrolled. Biopsie from metastatic lesions will be performed. A targeted cancer gene screen assay will be performed using DNA sequencing.

Results will be discussed during a molecular screening tumor board.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for all study procedures according to local regulatory requirements prior to enrollment into the study.
* Age ≥ 18 years.
* Histologically proven metastatic or locally recurrent CRC, NSCLC or melanoma.
* Tumor tissue (FFPE and frozen) from recurrent or metastatic lesions available for research purposes.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status >2.
* The biopsy procedure is estimated to be too risky for the patient.
* Any anti-VEGF or anti-VEGFR treatment administered less than 3 weeks before new biopsy procedure.
* No appropriate washout period for patients on anticoagulation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Quality of the biopsies | 1 month
  Percentage of frozen and FFPE core biopsies that are able to provide at least 1.5 μg of DNA of high quality suitable for molecular testing.
Technical failure rate. | 1 month
  Frequency of failures of each pathological and molecular tests.
Percentage of patients with results within the specified turnaround time | 1 month
  Percentage of patients for whom biopsy was performed within 10 working days from signature of the ICF and for whom all central laboratory results (pathology and molecular) will be available to the investigator within 15 working days from the time samples are received at the central laboratory (JBI).

SECONDARY OUTCOMES:
Feasibility of a tumor sequencing board. | 2 months
  Ability of the "tumor sequencing board" to assign patients to ongoing clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Aftimos, MD, Principal Investigator — Jules Bordet Insitute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium